CLINICAL TRIAL: NCT07230093
Title: The Effect of Combined Exercise Training on Physical Fitness Parameters in Children With Specific Learning Disabilities
Brief Title: Exercise and Physical Fitness in Children With Specific Learning Disabilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Meryem Sevim, PT, PhD, Lecturer, Department of Physiotherapy, Bartın Unıversity
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-SBB-0230
Record Dates: First submitted 2025-09-27; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Learning Disabilities
Keywords: Learning Disability; Physical Fitness; Combined Exercise; Children; Exercise Intervention
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups: the exercise group receives a combined exercise program for 8 weeks, 3 days per week, 45 minutes per session. The control group does not receive any intervention. Assessments of physical fitness parameters-including flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility-are performed before and after the intervention to evaluate changes.
Masking Description: No masking is applied in this study; participants, caregivers, and investigators are aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants receive a combined exercise program for 8 weeks, 3 days per week, 45 minutes per session. Physical fitness parameters-including flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility-are assessed before and after the intervention.
  Interventions: Behavioral: Combined Exercise Program
- Control Group (No Intervention): Participants do not receive any intervention. Physical fitness parameters-including flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility-are assessed at the same time points as the exercise group.

INTERVENTIONS:
Behavioral: Combined Exercise Program — Participants perform a combined exercise program for 8 weeks, 3 days per week, 45 minutes per session. Physical fitness parameters-including flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility-are assessed before and after the intervention. This program aims to improve gross and fine motor skills, balance, coordination, and overall physical fitness in children with specific learning difficulties.
  Arms: Exercise Group

SUMMARY:
Specific learning disabilities (SLD) are characterized by difficulties in reading, comprehension, arithmetic, and written expression, often accompanied by impairments in motor skills, balance, and coordination. However, physical difficulties in children with SLD are often overlooked in educational settings, and parental awareness of these issues remains limited.

This study aims to examine the effect of an 8-week combined exercise program-including balance, strength, and stretching exercises-on the physical fitness of children aged 7-14 years with SLD. Participants will be randomly assigned to either an exercise group or a control group.

The exercise intervention will be conducted three times per week for 45 minutes per session over eight weeks. Physical fitness will be evaluated through standardized field-based measures of balance, strength, flexibility, and endurance before and after the intervention. Data will be analyzed using SPSS 26.0, employing Wilcoxon, Mann-Whitney U, independent t-test, and paired t-test as appropriate.

The study is expected to emphasize the importance of physical activity for children with SLD and promote the inclusion of physiotherapy-based exercise programs in individualized support plans.

Primary Outcome Question: Does an 8-week combined exercise program improve balance, strength, flexibility, and endurance-key components of physical fitness-in children with specific learning disabilities compared to a control group?

DETAILED DESCRIPTION:
The term "Learning Disability" refers to difficulties in achieving expected academic performance in specific areas despite normal intelligence. In Turkey, learning disabilities encompass difficulties in one or more cognitive processes necessary for understanding and using language, either written or spoken. These difficulties may manifest in listening, speaking, reading, writing, spelling, attention, or mathematical operations.

Children with Specific Learning Disabilities (SLD) often experience not only academic difficulties but also deficits in motor skills, balance, and coordination. Physical fitness, defined as the ability to perform daily activities efficiently and safely, depends on multiple parameters including flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility. Regular exercise can improve these parameters, supporting children's physical, social, and cognitive development.

Despite the importance of physical fitness, studies on exercise interventions in SLD children are limited and mostly focus on balance. There is a lack of research investigating comprehensive combined exercise programs addressing multiple fitness components simultaneously.

The aim of this study is to examine the effects of a combined exercise program on physical fitness parameters in children with SLD aged 7-14 years. The primary objectives are:

To improve flexibility, muscular strength, muscular endurance, balance, coordination, speed, and agility.

To prevent deficits in gross and fine motor skills commonly observed in children with SLD.

To increase parental awareness of the importance of physical exercise in children with learning disabilities.

To provide a home-based exercise guide for children and parents to promote sustainable physical activity.

This randomized controlled study will be conducted in Bartın, Turkey, with 18 participants diagnosed with SLD according to official assessments. Participants will be randomly assigned to the exercise group, which will receive the combined exercise program, or to the control group, which will not receive intervention. Physical fitness parameters will be measured before and after the intervention to evaluate changes.

The combined exercise program consists of 8 weeks of progressive training, three times per week, 45 minutes per session, including warm-up, main exercise, and cool-down phases. Exercises target all major muscle groups and incorporate strength, flexibility, balance, coordination, speed, and agility components.

Hypothesis: H0: "Combined exercise training has a significant positive effect on the physical fitness parameters of children with SLD." The novelty of this study lies in addressing physical fitness comprehensively in SLD children, beyond academic interventions, and promoting sustainable exercise habits. Results are expected to contribute to both the scientific literature and practical guidance for education and rehabilitation programs for children with learning disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Exercise Group: Children aged 7-14 years diagnosed with Specific Learning Difficulty (SLD), with signed parental consent and child assent form
* Control Group: Children aged 7-14 years without SLD (healthy), with signed parental consent and child assent form

Exclusion Criteria:

* Children with physical disabilities preventing participation
* Children unable to cooperate with the assessments

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Balance Performance (Flamingo Balance Test) | Pre- and post-intervention (8 weeks)
  Description: Static balance will be assessed using the Flamingo Balance Test from the Eurofit Test Battery. Participants will stand on one leg on a narrow beam, and the number of falls within 1 minute will be recorded.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Number of falls (count)
  Interpretation: Lower scores indicate better balance.
Coordination Speed (Plate Tapping Test) | Before and after intervention (8 weeks)
  Description: Coordination and movement speed will be assessed using the Plate Tapping Test from the Eurofit Test Battery. The time required to complete 25 cycles of alternating taps will be recorded.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Seconds
  Interpretation: Lower scores indicate better performance.
Flexibility (Sit-and-Reach Test) | Before and after intervention (8 weeks)
  Description: Flexibility will be measured using the Sit and Reach Test, which assesses hamstring and lower back flexibility.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Centimeters
  Interpretation: Higher scores indicate greater flexibility.
Abdominal Muscle Endurance (Sit-Ups Test) | Before and after intervention (8 weeks)
  Description: Abdominal muscle endurance will be assessed using the Sit-Ups Test, recording the number of repetitions completed in 30 seconds.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Number of sit-ups (count)
  Interpretation: Higher scores indicate better endurance.
Lower Limb Power (Standing Long Jump Test) | Before and after intervention (8 weeks)
  Description: Explosive leg power will be evaluated using the Standing Long Jump Test. The best distance achieved in three trials will be recorded.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Centimeters
  Interpretation: Higher scores indicate better performance.
Cardiorespiratory Endurance (20 m Shuttle Run Test) | Before and after intervention (8 weeks)
  Description: Aerobic endurance will be assessed using the 20-meter Shuttle Run Test (Eurofit). The number of completed stages will be recorded.
  Time Frame: Baseline and 8 weeks
  Unit of Measure: Number of completed stages
  Interpretation: Higher scores indicate better endurance.
Age | Baseline (Pre-intervention)
  Measurement: Years
  Description: Chronological age of the participant will be recorded.
  Time Frame: Baseline (Pre-intervention)
Sex | Baseline (Pre-intervention)
  Measurement: Male / Female (categorical variable)
  Description: Biological sex will be recorded to explore potential differences in physical fitness outcomes.
  Time Frame: Baseline (Pre-intervention)
Body Mass Index (BMI) | Baseline (Pre-intervention)
  Measurement: kg/m²
  Description: BMI will be calculated using measured body weight and height (BMI = weight [kg] / height² [m²]). It will be used as a descriptive and covariate variable in analysis.
  Interpretation: Higher or lower BMI values will be examined in relation to physical fitness outcomes.
  Time Frame: Baseline (Pre-intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Vocational School of Health Services, Bartın, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No